CLINICAL TRIAL: NCT00572598
Title: Pilot Study of 18F Fluoropaclitaxel (FPAC) in Breast Cancer Patients and Normal Volunteers: Dosimetry and Imaging Feasibility
Brief Title: Pilot Study of 18F Fluoropaclitaxel (FPAC)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HM03748
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: PET; multidrug resistance; fluoropaclitaxel; paclitaxel; breast cancer; dosimetry; imaging feasibility
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 4- [F-18] fluoropaclitaxel — 4- [F-18] fluoropaclitaxel, <84 micrograms, <10 mCi, IV followed by PET/CT imaging
  Other Names: FPAC

SUMMARY:
Multidrug resistance (MDR) is a cause of treatment failure in many cancer patients. MDR refers to a phenotype whereby a tumor is resistant to a large number of natural chemotherapeutic drugs. Having prior knowledge of the presence of such resistance would decrease morbidity from unsuccessful therapy and allow for the selection of individuals who may benefit from co-administration of MDR inhibiting drugs. The Tc-99m labeled single photon emitting radiotracers sestamibi and tetrofosmin have shown some predictive value. However, positron-emitting (PET) radiotracers, which allow for dynamic, quantitative imaging, hold the promise of more accurate and specific identification of MDR tumors.

Objective:

To obtain human safety data, to demonstrate imaging feasibility with FPAC, to obtain human biodistribution and to obtain preliminary evidence of breast tumor uptake concordance with response to therapy.

DETAILED DESCRIPTION:
18F flouropaclitaxel (FPAC) distribution in malignant tumors is expected to be similar to that of paclitaxel. It is proposed that by monitoring the influx and efflux of FPAC in vivo using PET imaging, we will be able to determine if a tumor retains the drug (is drug sensitive) or pumps it out (is drug resistant). The efflux rate of FPAC in the tumor should be proportional the amount of Pgp present and therefore should be a predictor of treatment failure. If this method is successful at identifying MDR, patients can be spared a course of ineffective chemotherapy and can be started on alternative drugs or, if available, an effective MDR modulator can be administered prior to treatment.

In order to validate the biodistribution in non-human primate, 3 normal volunteers will be recruited to participate in a dosimetry PET imaging protocol.

Often, patients with breast cancer are treated with chemotherapy prior to definitive surgical removal of the primary tumor. Three patients with breast cancer who are candidates for this neoadjuvant chemotherapy will also be recruited to participate in this study, in order to demonstrate the feasibility of tumor imaging. As these patients will be receiving chemotherapy (likely paclitaxel), a preliminary correlation with FPAC uptake and tumor response can also be attempted in this pilot study.

Primary Objective

--To obtain human dosimetry and monitor for potential physiologic effects following 4-[F-18] fluoropaclitaxel (FPAC) administration

Secondary Objectives

* a.To characterize tracer uptake in tumors and normal tissues and develop robust methods for analysis of FPAC kinetics in breast tumors
* b.To optimize the imaging protocol for FPAC, and, if feasible, reduce to 1 or 2 static scans

ELIGIBILITY:
Normal Volunteers

Inclusion Criteria:

* Subjects must be 18 years or older for inclusion in this study. Because no dosing or adverse event data are currently available on the use of FPAC in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.

  * All subjects must sign a written informed consent document and a Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines.
  * If female, the subject must be postmenopausal for a minimum of one year, or surgically sterile, or be within 14 days of onset of a menstrual period or have a negative beta human chorionic gonadotropin (ßHCG) blood test.
  * Subjects must have normal organ and marrow function as defined below:
  * Leukocytes >3,000/μL
  * absolute neutrophil count >1,500/μL
  * platelets >100,000/μL
  * total bilirubin within normal institutional limits
  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <= 2.5 times the institutional upper limit of normal
  * Creatinine within normal institutional limits OR, in subjects with creatinine levels above institutional normal, creatinine clearance >60 mL/min/1.73 m2

Exclusion Criteria:

* Subject with a known bleeding disorder

  * Subjects who have received chemotherapy within 1 year of entry into study
  * Subjects with a history of liver or kidney disease
  * Subjects who are receiving any other investigational agents
  * Subjects having severe claustrophobia or other condition that would make them unable to lie still for the duration of the study
  * Subjects with immunodeficiencies that predispose a subject to specific or non-specific mediator release
  * Subjects with uncontrolled intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
  * Subjects who are pregnant or lactating or who suspect they might be pregnant. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with FPAC, breastfeeding should be discontinued if the mother receives FPAC.

Breast Cancer Patients

Inclusion Criteria:

* Subjects must have a history of histologically or cytologically confirmed breast cancer with estimated lesion size of >1cm.

  * Subjects must be 18 years or older for inclusion in this study. Because no dosing or adverse event data are currently available on the use of FPAC in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
  * All subjects must sign a written informed consent document and a HIPAA authorization in accordance with institutional guidelines.
  * If female, the subject must be postmenopausal for a minimum of one year, be surgically sterile, be within 14 days of onset of a menstrual period, or have a negative ßHCG blood test.
  * Subjects must have normal organ and marrow function as defined below:
  * Leukocytes >3,000/μL
  * absolute neutrophil count >1,500/μL
  * platelets >100,000/μL
  * total bilirubin within normal institutional limits
  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <= 2.5 times the institutional upper limit of normal
  * Creatinine within normal institutional limits OR, in subjects with creatinine levels above institutional normal, creatinine clearance >60 mL/min/1.73 m2

Exclusion Criteria:

•as above

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Imaging feasibility and dosimetry | <6months

CONTACTS AND LOCATIONS:
Overall Officials: Harry D. Bear, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Kalen JD, Hirsch JI, Kurdziel KA, Eckelman WC, Kiesewetter DO. Automated synthesis of 18F analogue of paclitaxel (PAC): [18F]Paclitaxel (FPAC). Appl Radiat Isot. 2007 Jun;65(6):696-700. doi: 10.1016/j.apradiso.2006.10.015. Epub 2006 Dec 11. PMID 17161952
- [Result] Kurdziel KA, Kalen JD, Hirsch JI, Wilson JD, Agarwal R, Barrett D, Bear HD, McCumiskey JF. Imaging multidrug resistance with 4-[18F]fluoropaclitaxel. Nucl Med Biol. 2007 Oct;34(7):823-31. doi: 10.1016/j.nucmedbio.2007.04.011. Epub 2007 Jul 5. PMID 17921033
- [Result] Kurdziel KA, Kalen JD, Hirsch JI, Wilson JD, Bear HD, Logan J, McCumisky J, Moorman-Sykes K, Adler S, Choyke PL. Human dosimetry and preliminary tumor distribution of 18F-fluoropaclitaxel in healthy volunteers and newly diagnosed breast cancer patients using PET/CT. J Nucl Med. 2011 Sep;52(9):1339-45. doi: 10.2967/jnumed.111.091587. Epub 2011 Aug 17. PMID 21849404
- See also: VCU Molecular Imaging Center Home Page — http://www.molecularimaging.vcu.edu